CLINICAL TRIAL: NCT03241498
Title: GP Practice Based Pharmacist Input to Medicines Optimisation
Brief Title: General Practitioner (GP) Practice Based Pharmacist Input to Medicines Optimisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Medicines Optimisation Innovation Centre (MOIC) (Unknown); Association of the British Pharmaceutical Industry (ABPI) (Unknown)
Responsible Party: Principal Investigator, James McElnay, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: QUB B16/46
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Medication Adherence
Keywords: Medicines optimisation; Healthcare resource utilisation; HRQOL; Pharmacist-led; GP based
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: A prospective, multi-centre, randomised intervention study will be conducted simultaneously in four different regions of the United Kingdom (UK), namely:
  1. Northern Health and Social Care Trust (NHSCT) and Western Health and Social Care Trust (WHSCT), Northern Ireland
  2. North West Coast Academic Health Science Network (AHSN), England
  3. Wessex AHSN, England
  4. Eastern AHSN, England
  Two GP practices will participate in the research in each of these four geographical areas. The pragmatic sample size at each site will be 50 intervention patients and 50 control patients completing a six month follow-up period i.e. a total of 800 patients (400 intervention and 400 control patients) across the eight participating GP practices. An over-recruitment of 20%, i.e. 60 each of both control and interventions patients per practice, will be recruited into the study to take account of patients who drop out of the study and/or are lost to follow up.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): All patients allocated to the control group, who on checking meet the study entry criteria and who consent (written informed consent) to participate in the research, will be asked to complete the three study questionnaires (see below) and will be advised that repeat questionnaires will be distributed by post at the end of the study (6 months) for completion at home and return by post. The patients will continue to receive all services provided by the GP practice (normal care) but will not receive the bespoke clinical pharmacist intervention which is being evaluated in this research study.
- Intervention arm (Experimental): Participants meeting all study entry criteria who are allocated to the intervention group will also be asked to complete the three study questionnaires. Having completed the questionnaires they will receive the medicines optimisation intervention by the clinical pharmacist. They will be asked to return for repeat appointments with the clinical pharmacist at 2 and 4 months and will be advised that they will be asked to complete the study questionnaires again at the end of the study (at home, via post at 6 months).
  Interventions: Other: Medicines optimisation

INTERVENTIONS:
Other: Medicines optimisation
  Arms: Intervention arm

SUMMARY:
The study is a United Kingdom (UK) based multi-centre study which will evaluate the impact of a medication optimisation intervention (delivered in GP practices by pharmacists to patients at risk of medication related problems), on healthcare resource utilisation and patient outcomes. Pharmacists in 4 areas across the UK (3 in England and 1 in Northern Ireland) will engage with patients, thought to be at a higher risk of medication related problems, within their GP practice in order to help identify areas for improvement

DETAILED DESCRIPTION:
Drug therapy is growing more complex as patients increasingly suffer from a number of co-morbidities. Accordingly, in clinical medicine, a wide range of medication related problems may arise (1). A medication related problem (MRP) is defined as "an event or circumstance involving drug therapy that actually or potentially interferes with desired health outcomes" (2). These problems have been found to lead to more hospital admissions and thus increase the cost of healthcare provision (3, 4). For instance, Winterstein et al. carried out a meta-analysis of research in this area which showed that 7.1% of hospital admissions were attributable to a drug related problem, of which 59% appeared avoidable (5). Moreover, a large study in the United Kingdom showed that these admissions cost the National Health Service (NHS) up to £466 million annually, which is 0.59% of the British health care budget (6).

Medication related problems (MRPs) remain a serious concern particularly in primary care settings. A recent UK study found that one in 20 prescription items in general practice included an error, affecting 1 in 8 patients. Although the majority of these errors were described as being either mild or moderate in severity, 1 in 550 of all prescription items contained an error determined to be severe (7). In addition, significant medication wastage has been found within general practice settings in England with an estimated £300 million worth of prescribed medications being wasted each year in primary and community care (8). Optimisation of drug therapy and prevention of MRPs can reduce health care expenditure, potentially save lives and enhance patient quality of life (9-13).

Medicines optimisation is defined as 'a person-centred approach to safe and effective medicines use, to ensure people obtain the best possible outcomes from their medicines. Medicines optimisation applies to people who may or may not take their medicines effectively. Shared decision-making is an essential part of evidence-based medicine, seeking to use the best available evidence to guide decisions about the care of the individual patient, taking into account their needs, preferences and values' (14, 15, 16).

Medicines optimisation requires more patient engagement and professional collaboration within health and social care settings. It focuses on actions taken by all health and social care practitioners. To support the medicines optimisation agenda a guide on medicines optimisation has been produced by The Royal Pharmaceutical Society (RPS) the aim of which is to help patients make the most of their medicines (17). This guide involves four key principles for medicines optimisation in order to achieve improved patient outcomes (16). These principles are as follows:

(i) Aim to understand the patient's experience (ii) Evidence based choice of medicines (iii) Ensure medicines use is as safe as possible (iv) Make medicines optimisation part of routine practice

In order to support the implementation of the guiding principles, NHS England launched the prototype medicines optimisation dashboard in 2014. The dashboard aims to 'encourage Clinical Commissioning Groups (CCGs) and healthcare Trusts to think more about how well their patients are supported to use medicines and less about focusing on cost and volume of drugs' (16).

Primary care systems have started utilising a team based approach to care delivery. Pharmacists have been increasingly recognised as a part of the healthcare professional team within primary care settings in many countries (18). This integration of pharmacists into primary health care systems was found to have significant benefits that included reduction of errors, effective identification and resolution of medication related problems, improvements in medication adherence, improved patient outcomes, relief of work pressure on GPs, improved communication and cooperation between health professionals, and strengthened team working within primary care (18-22).

Despite the expansion of the role of pharmacists in the primary health care setting, limited research has been conducted to evaluate the impact of pharmacist input on health service utilisation and cost.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if they have any of the following:

* Have had at least 1 unplanned hospital admission or 2 or more accident and emergency department (A&E) attendances in the previous 12 months.
* Prescribed ≥ 6 regular oral/systemic, long term medicines.
* Has ≥ 2 long-term chronic conditions.

Exclusion Criteria:

* Patient is residing in a nursing home or a care home.
* Patient is considered unable to give written informed consent e.g. Alzheimer's disease.
* Palliative care patients.
* Patient has had ≥ 4 unplanned admissions to hospital in the previous 6 months.
* Patient is participating in another intervention research project within the practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Number of unplanned hospital admissions | Recruitment - 6 months post intervention
  Number of unplanned admissions to hospital over the follow-up period will be collected for both control and intervention patients
Number of A&E attendances | Recruitment - 6 months post intervention
  Number of attendance to the A&E department over the follow-up period will be collected for both control and intervention patients
Number of GP consultations | Recruitment - 6 months post intervention
  Number of unplanned consultations with the patient's GP over the follow-up period will be collected for both control and intervention patients

SECONDARY OUTCOMES:
Medication appropriateness index (MAI) score | Recruitment - 6 months post intervention
  MAI scores will be calculated at the beginning and end of the project for each patient recruited into the study
Number of medication related problems | Recruitment - 6 months post intervention
  Number of medication related problems will be calculated at the beginning and end of the project for each patient recruited into the study
Health-related quality of life (HRQOL) | Recruitment - 6 months post intervention
  HRQOL scores will be calculated using the EQ-5D tool at the beginning and end of the project for each patient recruited into the study
Medication Adherence report scale (MARS) | Recruitment - 6 months post intervention
  MARS scores will be calculated at the beginning and end of the project for each patient recruited into the study
Beliefs about medicines questionnaire (BMQ) | Recruitment - 6 months post intervention
  BMQ scores will be calculated at the beginning and end of the project for each patient recruited into the study
Patient satisfaction with GP services | Recruitment - 6 months post intervention
  Patients will be asked to complete a bespoke satisfaction questionnaire in order to assess their satisfaction with the new service which has been provided
Patient laboratory data relevant to medications being received | Recruitment - 6 months post intervention
  Pertinent laboratory data will be collected throughout the intervention period and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: James C McElnay, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Northern Health and Social Care Trust, Antrim, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Final results will be disseminated through relevant academic press

REFERENCES:
- [Derived] Syafhan NF, Al Azzam S, Williams SD, Wilson W, Brady J, Lawrence P, McCrudden M, Ahmed M, Scott MG, Fleming G, Hogg A, Scullin C, Horne R, Ahir H, McElnay JC. General practitioner practice-based pharmacist input to medicines optimisation in the UK: pragmatic, multicenter, randomised, controlled trial. J Pharm Policy Pract. 2021 Jan 4;14(1):4. doi: 10.1186/s40545-020-00279-3. PMID 33397509